CLINICAL TRIAL: NCT02414633
Title: Special Investigation (Working Productivity and Activity Impairment in Japanese Patients With Psoriatic Arthritis)
Brief Title: Special Investigation in Patients With Psoriatic Arthritis (PsA) (Working Productivity and Activity Impairment [WPAI])
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-084
Record Dates: First submitted 2015-01-30; First posted 2015-04-13 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Humira: Subjects with Psoriatic Arthritis taking adalimumab under conditions of daily clinical practice.

SUMMARY:
A special investigation (post marketing observational study [PMOS]/non-mandatory) of HUMIRA® in Japanese psoriatic arthritis patients who are engaged in paid work.

ELIGIBILITY:
Inclusion Criteria:

* Paid workers (including part-time) with Psoriatic Arthritis, who have never administered adalimumab, and are diagnosed by ClASsification of Psoriatic ARthritis (CASPAR) criteria

Exclusion Criteria:

* Subjects showing decreased basic activities of daily life such as hospitalization and bedridden
* Subjects with contraindications to adalimumab

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-arm, multi-center study with a prospective cohort.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Kurimoto, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Nakagawa H, Tanaka Y, Sano S, Kameda H, Taniguchi A, Kashiwagi T, Kawaberi T, Kimura J, Morita A. Real-World Postmarketing Study of the Impact of Adalimumab Treatment on Work Productivity and Activity Impairment in Patients with Psoriatic Arthritis. Adv Ther. 2019 Mar;36(3):691-707. doi: 10.1007/s12325-018-0866-y. Epub 2019 Jan 19. PMID 30661197
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Humira
Started | 148
Completed | 148
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Humira
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Work Productivity and Activity Impairment Psoriatic Arthritis Questionnaire (WPAI:PsA) Percentage of Overall Work Impairment (OWI): Change From Baseline to Week 24
Description: WPAI:PsA is a questionnaire used to evaluate lost productivity due to PsA; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Percentage of overall work impairment due to PsA (OWI) is calculated as: Absenteeism + (1 - Absenteeism) * Presenteeism. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 24
Population: Efficacy analysis population: All enrolled participants with available OWI scores.
Measure: Mean (Standard Deviation); unit: percentage of OWI
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of OWI
  Baseline | 40.22 (32.84)
  Change from Baseline to Week 24: number analyzed (Participants) | 79
  Change from Baseline to Week 24 | -25.24 (35.27)

2. Secondary Outcome: WPAI:PsA Percentage of OWI: Change From Baseline to Weeks 4, 12, and 16
Description: as for outcome 1
Time Frame: Baseline (Week 0), Week 4, Week 12, and Week 16
Population: Efficacy analysis population: All enrolled participants with available OWI scores.
Measure: Mean (Standard Deviation); unit: percentage of OWI
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of OWI
  Baseline | 40.22 (32.84)
  Change from Baseline to Week 4: number analyzed (Participants) | 70
  Change from Baseline to Week 4 | -16.35 (24.35)
  Change from Baseline to Week 12: number analyzed (Participants) | 69
  Change from Baseline to Week 12 | -18.83 (32.64)
  Change from Baseline to Week 16: number analyzed (Participants) | 64
  Change from Baseline to Week 16 | -25.91 (32.26)

3. Secondary Outcome: WPAI:PsA Absenteeism: Change From Baseline to Weeks 4, 12, 16 and 24
Description: WPAI:PsA is a questionnaire used to evaluate lost productivity due to PsA; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Absenteeism (percentage of work time missed due to PsA) is calculated as the number of hours of work missed due to PsA / (number of hours of work missed due to PsA + number of hours worked) * 100. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of work time missed
  Baseline | 8.41 (22.97)
  Change from Baseline to Week 4: number analyzed (Participants) | 70
  Change from Baseline to Week 4 | -5.13 (16.96)
  Change from Baseline to Week 12: number analyzed (Participants) | 69
  Change from Baseline to Week 12 | -4.96 (16.73)
  Change from Baseline to Week 16: number analyzed (Participants) | 64
  Change from Baseline to Week 16 | -5.37 (17.54)
  Change from Baseline to Week 24: number analyzed (Participants) | 79
  Change from Baseline to Week 24 | -4.90 (20.13)

4. Secondary Outcome: WPAI:PsA Presenteeism: Change From Baseline to Weeks 4, 12, 16 and 24
Description: WPAI:PsA is a questionnaire used to evaluate lost productivity due to PsA; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Presenteeism (percentage of impairment while working due to PsA) is calculated as the patient's rating of how much PsA affected productivity while working (0 = no effect; 10 = completely prevented from working) / 10 * 100. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of impairment while working
  Baseline | 37.5 (32.0)
  Change from Baseline to Week 4: number analyzed (Participants) | 74
  Change from Baseline to Week 4 | -15.1 (24.3)
  Change from Baseline to Week 12: number analyzed (Participants) | 73
  Change from Baseline to Week 12 | -16.2 (31.1)
  Change from Baseline to Week 16: number analyzed (Participants) | 67
  Change from Baseline to Week 16 | -24.9 (31.5)
  Change from Baseline to Week 24: number analyzed (Participants) | 82
  Change from Baseline to Week 24 | -24.3 (33.4)

5. Secondary Outcome: WPAI:PsA Activity Impairment: Change From Baseline to Weeks 4, 12, 16 and 24
Description: WPAI:PsA is a questionnaire used to evaluate lost productivity due to PsA; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Activity impairment (percentage of activity impairment due to PsA) is calculated as the patient's rating of how much PsA affected their ability to do regular daily activities, other than working at a job (0 = no effect; 10 = completely prevented from working) / 10 * 100. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Humira
Number analyzed (Participants) | 104
percentage of impairment
  Baseline | 41.7 (30.1)
  Change from Baseline to Week 4: number analyzed (Participants) | 72
  Change from Baseline to Week 4 | -17.4 (23.0)
  Change from Baseline to Week 12: number analyzed (Participants) | 73
  Change from Baseline to Week 12 | -20.1 (28.5)
  Change from Baseline to Week 16: number analyzed (Participants) | 66
  Change from Baseline to Week 16 | -25.0 (32.0)
  Change from Baseline to Week 24: number analyzed (Participants) | 82
  Change from Baseline to Week 24 | -27.1 (32.7)

6. Secondary Outcome: Psoriatic Arthritis Screening and Evaluation Questionnaire (PASE): Change From Baseline to Weeks 4, 12, 16 and 24
Description: The PASE is a patient-administered questionnaire used to screen patients with psoriasis for evidence of psoriatic arthritis. The PASE consists of 15 questions divided into 2 subscales (system sub-scale and function sub-scale); 7 questions assess symptoms and 8 questions assess function. Questions are scored on a numeric scale ranging from 1 (strongly disagree) to 5 (strongly agree), with a total possible PASE score of 15 to 75. Individuals who are more likely to have PsA will score higher than individuals without PsA. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 106
units on a scale
  Baseline | 47.4 (11.7)
  Change from Baseline to Week 4: number analyzed (Participants) | 74
  Change from Baseline to Week 4 | -11.8 (11.0)
  Change from Baseline to Week 12: number analyzed (Participants) | 75
  Change from Baseline to Week 12 | -14.5 (13.8)
  Change from Baseline to Week 16: number analyzed (Participants) | 67
  Change from Baseline to Week 16 | -16.6 (13.6)
  Change from Baseline to Week 24: number analyzed (Participants) | 83
  Change from Baseline to Week 24 | -18.1 (14.0)

7. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score: Change From Baseline to Weeks 4, 12, 16 and 24
Description: PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on of the lesions rated on a a scale from 0 (no symptoms) to 4 (very marked), together with the percentage of the area affected, rated on a scale from 0 (0%) to 6 (100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 98
units on a scale
  Baseline | 8.97 (8.55)
  Change from Baseline to Week 4: number analyzed (Participants) | 67
  Change from Baseline to Week 4 | -4.06 (5.46)
  Change from Baseline to Week 12: number analyzed (Participants) | 73
  Change from Baseline to Week 12 | -5.14 (6.49)
  Change from Baseline to Week 16: number analyzed (Participants) | 61
  Change from Baseline to Week 16 | -7.35 (7.92)
  Change from Baseline to Week 24: number analyzed (Participants) | 77
  Change from Baseline to Week 24 | -6.63 (6.72)

8. Secondary Outcome: Disease Activity Score 28, C-reactive Protein (DAS28 [CRP]): Change From Baseline to Weeks 4, 12, 16 and 24
Description: DAS28 (CRP) is calculated using the number of tender and swollen joints (out of 28 counted), C-reactive protein (CRP) level, and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0 to 10. A score less than 2.6 indicates clinical remission, a score of 2.6 to 3.2 indicates low disease activity, a score of 3.2 to less than 5.1 indicates moderate disease activity, and a score of 5.1 or greater indicates high disease activity. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 61
units on a scale
  Baseline | 3.77 (1.33)
  Change from Baseline to Week 4: number analyzed (Participants) | 28
  Change from Baseline to Week 4 | -1.48 (0.86)
  Change from Baseline to Week 12: number analyzed (Participants) | 29
  Change from Baseline to Week 12 | -1.83 (0.92)
  Change from Baseline to Week 16: number analyzed (Participants) | 27
  Change from Baseline to Week 16 | -1.84 (1.07)
  Change from Baseline to Week 24: number analyzed (Participants) | 26
  Change from Baseline to Week 24 | -2.13 (1.20)

9. Secondary Outcome: Disease Activity Score 28, Erythrocyte Sedimentation Rate (DAS28 [ESR]): Change From Baseline to Weeks 4, 12, 16 and 24
Description: DAS28 (ESR) is calculated using the number of tender and swollen joints (out of 28 counted), erythrocyte sedimentation rate (ESR), and the patient's global assessment of disease activity via the visual analog scale (VAS). The calculated range of DAS28-4 is 0 to 10. A score less than 2.6 indicates clinical remission, a score of 2.6 to 3.2 indicates low disease activity, a score of 3.2 to less than 5.1 indicates moderate disease activity, and a score of 5.1 or greater indicates high disease activity. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 48
units on a scale
  Baseline | 4.25 (1.40)
  Change from Baseline to Week 4: number analyzed (Participants) | 19
  Change from Baseline to Week 4 | -1.60 (0.65)
  Change from Baseline to Week 12: number analyzed (Participants) | 22
  Change from Baseline to Week 12 | -1.99 (0.92)
  Change from Baseline to Week 16: number analyzed (Participants) | 21
  Change from Baseline to Week 16 | -2.13 (0.94)
  Change from Baseline to Week 24: number analyzed (Participants) | 20
  Change from Baseline to Week 24 | -2.57 (1.20)

10. Secondary Outcome: Tender Joint Count (TJC68): Change From Baseline to Weeks 4, 12, 16 and 24
Description: At each study visit, a joint evaluator assessed whether a particular joint was "tender or painful" where presence of tenderness was scored as "1" and the absence of tenderness was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. The total TJC68, which is based on 68 joints, was derived as the sum of all "1s" thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for TJC68 was 0 to 68, with a higher score indication a greater degree of tenderness. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Humira
Number analyzed (Participants) | 99
tender joints
  Baseline | 7.2 (8.7)
  Change from Baseline to Week 4: number analyzed (Participants) | 64
  Change from Baseline to Week 4 | -3.8 (7.2)
  Change from Baseline to Week 12: number analyzed (Participants) | 73
  Change from Baseline to Week 12 | -4.8 (9.7)
  Change from Baseline to Week 16: number analyzed (Participants) | 60
  Change from Baseline to Week 16 | -4.5 (7.3)
  Change from Baseline to Week 24: number analyzed (Participants) | 75
  Change from Baseline to Week 24 | -6.2 (9.4)

11. Secondary Outcome: Swollen Joint Count (SJC66): Change From Baseline to Weeks 4, 12, 16 and 24
Description: At each study visit, a joint evaluator assessed whether a particular joint was swollen where presence of swelling was scored as "1" and the absence of swelling was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. The total SJC66, which is based on 66 joints, was derived as the sum of all "1s" thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for SJC66 was 0 to 66, with a higher score indicating a greater degree of swelling. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 16, and 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Humira
Number analyzed (Participants) | 99
swollen joints
  Baseline | 5.3 (7.0)
  Change from Baseline to Week 4: number analyzed (Participants) | 64
  Change from Baseline to Week 4 | -2.7 (5.0)
  Change from Baseline to Week 12: number analyzed (Participants) | 73
  Change from Baseline to Week 12 | -3.9 (6.6)
  Change from Baseline to Week 16: number analyzed (Participants) | 60
  Change from Baseline to Week 16 | -3.9 (5.4)
  Change from Baseline to Week 24: number analyzed (Participants) | 75
  Change from Baseline to Week 24 | -4.9 (7.2)

12. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): Change From Baseline to Weeks 12 and 24
Description: The BASDAI uses a scale from 1 (no problem) to 10 (worst problem) to answer 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain/swelling, areas of localized tenderness (also called enthesitis, or inflammation of tendons and ligaments), morning stiffness duration, and morning stiffness severity. To give each symptom equal weighting, the mean (average) of the two scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final BASDAI score ranging from 0-10. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 12, and Week 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 99
units on a scale
  Baseline | 4.203 (2.334)
  Change from Baseline to Week 12: number analyzed (Participants) | 50
  Change from Baseline to Week 12 | -2.058 (2.212)
  Change from Baseline to Week 24: number analyzed (Participants) | 64
  Change from Baseline to Week 24 | -2.745 (2.573)

13. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI): Change From Baseline to Weeks 12 and 24
Description: The HAQ-DI is a patient-reported outcome which is usually self-administered by the patient. The HAQ-DI assesses the categories of dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. The patients report the amount of difficulty they have in performing these activities using a scale ranging from 0 (can be performed without any difficulty) to 3 (cannot be done at all). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability. Change from baseline was calculated as the value at baseline minus the value at each subsequent time point. A negative change represents improvement.
Time Frame: Baseline (Week 0), Week 12, and Week 24
Population: Efficacy analysis population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 105
units on a scale
  Baseline | 0.5429 (0.5017)
  Change from Baseline to Week 12: number analyzed (Participants) | 57
  Change from Baseline to Week 12 | -0.2522 (0.4255)
  Change from Baseline to Week 24: number analyzed (Participants) | 66
  Change from Baseline to Week 24 | -0.3996 (0.4719)

14. Secondary Outcome: Enthesitis: Change From Baseline to Final Visit
Description: The percentage of participants with enthesitis.
Time Frame: Baseline (Week 0) and final visit (up to 24 weeks)
Population: Efficacy analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of participants
  Baseline | 36.8
  Final Visit | 12.3

15. Secondary Outcome: Dactylitis: Change From Baseline to Final Visit
Description: The percentage of participants with dactylitis.
Time Frame: Baseline (Week 0) and final visit (up to 24 weeks)
Population: Efficacy analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of participants
  Baseline | 55.7
  Final Visit | 7.5

16. Secondary Outcome: Spondylitis: Change From Baseline to Final Visit
Description: The percentage of participants with spondylitis.
Time Frame: Baseline (Week 0) and final visit (up to 24 weeks)
Population: Efficacy analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of participants
  Baseline | 29.2
  Final Visit | 4.7

17. Secondary Outcome: Nail Psoriasis: Change From Baseline to Final Visit
Description: The percentage of participants with nail psoriasis .
Time Frame: Baseline (Week 0) and final visit (up to 24 weeks)
Population: Efficacy analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 106
percentage of participants
  Baseline | 50.9
  Final Visit | 29.2

18. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probable, possible, not related, or impossible to judge. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the physician obtained the patient's authorization or informed consent until the end of the study (week 28 or discontinuation).
Time Frame: From the first dose of study drug until the end of the study (up to 24 weeks)
Population: Safety analysis population: All participants enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 148
participants
  Any TEAE | 28
  Any TESAE | 4

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until the end of the study (up to 24 weeks)]
Arm/Group | Humira
All-Cause Mortality (participants affected / at risk) | 0/148
Serious Adverse Events (participants affected / at risk) | 4/148
Other Adverse Events (participants affected / at risk) | 28/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=148)
Cellulitis staphylococcal (Infections and infestations) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lupus nephritis (Renal and urinary disorders) | 1
Paradoxical drug reaction (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=148)
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 3
Herpes zoster infection neurological (Infections and infestations) | 1
Hypoaesthesia (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Injection site erythema (General disorders) | 1
Injection site pruritus (General disorders) | 1
Oedema (General disorders) | 1
Paradoxical drug reaction (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Antinuclear antibody positive (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Cell marker increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02414633/Prot_SAP_000.pdf